CLINICAL TRIAL: NCT04075292
Title: A Randomized, Multicenter, Open-Label, Phase 3 Study to Evaluate the Efficacy and Safety of Acalabrutinib Versus Chlorambucil Plus Rituximab in Subjects With Previously Untreated Chronic Lymphocytic Leukemia
Brief Title: Study of Acalabrutinib Versus Chlorambucil Plus Rituximab in Adult Subjects With Previously Untreated Chronic Lymphocytic Leukemia
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D822BC00001
Record Dates: First submitted 2019-08-19; First posted 2019-08-30 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Untreated Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; Acalabrutinib; Progression-free Survival
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — acalabrutinib; Rituximab; Chlorambucil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acalabrutinib (Experimental): Acalabrutinib will be orally administered until disease progression or unacceptable toxicity
  Interventions: Drug: Acalabrutinib
- Rituximab and Chlorambucil (Active Comparator): Chlorambucil orally administered and Rituximab via IV infusion for 6 cycles
  Interventions: Drug: Rituximab; Drug: Chlorambucil

INTERVENTIONS:
Drug: Acalabrutinib — acalabrutinib 100 mg twice daily orally
  Arms: Acalabrutinib
Drug: Rituximab — Rituximab: 375 mg/m2 IV infusion on Day 1 of Cycle 1. 500 mg/m2 IV infusion on Day 1 for each of subsequent cycles (Cycles 2-6)
  Arms: Rituximab and Chlorambucil
Drug: Chlorambucil — Chlorambucil: 0.5 mg/kg body weight orally on Day 1 and Day 15 of Cycles 1-6
  Arms: Rituximab and Chlorambucil

SUMMARY:
This is a randomized, multicenter, open-label, Phase 3 study to evaluate the efficacy and safety of Acalabrutinib versus Chlorambucil plus Rituximab in subjects with Previously Untreated Chronic Lymphocytic Leukemia.

DETAILED DESCRIPTION:
Patients be randomized in a 1:1 ratio into 2 arms to receive either acalabrutinib monotherapy (Arm A) or rituximab in combination with chlorambucil (Arm B). The primary objective of this study is to compare the efficacy of acalabrutinib relative to chlorambucil plus rituximab in subjects with previously untreated chronic lymphocytic leukemia without del(17p) or TP53 mutation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women: (a) ≥65 years of age OR (b) >18 and <65 years of age, provided that they meet at least one of the following criteria: (i) Creatinine clearance 30 to 69 mL/min using the Cockcroft-Gault equation (iwCLL guidelines) (ii) A score higher than 6 on the Cumulative Illness Rating Score-Geriatric (CIRS G)
* ECOG performance status of 0, 1, or 2
* Diagnosis of CLL that meets published diagnostic criteria (Hallek 2018)
* Active disease per IWCLL 2018 criteria that requires treatment
* Adequate bone marrow function
* Adequate renal and hepatic function

Exclusion Criteria:

* Known detected del(17p) or TP53 mutation
* Transformation of CLL to aggressive non-Hodgkin lymphoma (NHL) (eg, Richter's transformation, PLL, or diffuse large B cell lymphoma [DLBCL]), or central nervous system (CNS) involvement by leukemia
* History of prior malignancy except for the following: (a) Curatively treated basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix at any time prior to study (b) Other cancers not specified above which have been curatively treated by surgery and/or radiation therapy from which subject is disease-free for ≥3 years without further treatment
* Significant cardiovascular disease
* Known history of infection with human immunodeficiency virus (HIV)
* Serologic status reflecting active hepatitis B or C infection
* Any active systemic infection (eg, bacterial, viral, or fungal infection) requiring systemic treatment
* History of stroke or intracranial hemorrhage within 6 months before first dose of study drug
* Major surgical procedure within 30 days of first dose of study drug
* Any prior CLL-specific therapies
* Corticosteroid use >20 mg within 1 week before first dose of study drug, except as indicated for other medical conditions
* Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists
* For women only: breastfeeding or pregnant

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2027-01-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Lugui Qiu, MD, Principal Investigator — Chinese Academy of Medical Science Affiliated Hospital of Hematology
Locations (37):
- China (19):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Changzhou
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shijiazhuang
  - Research Site, Suzhou
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Xuzhou
  - Research Site, Zhengzhou
- Philippines (6):
  - Research Site, Baguio City
  - Research Site, Cebu
  - Research Site, Davao City
  - Research Site, Makati
  - Research Site, Manila
  - Research Site, Quezon City
- Taiwan (6):
  - Research Site, Chiayi City
  - Research Site, Hualien City
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D822BC00001&attachmentIdentifier=88da95ab-439d-4f9d-bb83-80f1c40de09a&fileName=d822bc00001-CSR_Synopsis_Final_Redacted_PDFA.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D822BC00001&attachmentIdentifier=77cbdb95-97df-41c5-89a6-7e00bae22137&fileName=d822bc00001-csp-v5_Final_Redacted_PDFA.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D822BC00001&attachmentIdentifier=fa0e164e-6df4-43a5-aff9-a564fd635052&fileName=D822bc00001-sap-ed-2.0_19Dec2023_Final_Redacted_PDFA.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase III, multicenter, randomized, open-label study was conducted in participants with previously untreated chronic lymphocytic leukemia (CLL) without del(17p) or TP53 mutation at 46 sites across 5 countries. Results are presented up to data cut-off (DCO) date of 03 January 2024.
Pre-assignment Details: A total of 155 participants were randomized in 1:1 ratio to acalabrutinib treatment arm or chlorambucil plus rituximab treatment arm. All participants should receive the same dose within their respective treatment arms.
Groups:
- Acalabrutinib: Participants received acalabrutinib 100 milligram (mg) orally twice daily (BID) in 28-day cycles until progression of disease (PD) or any other treatment discontinuation criterion was met.
- Chlorambucil Plus Rituximab: Participants received chlorambucil 0.5 milligram per kilogram (mg/kg) body weight orally on Day 1 and Day 15 of all 28-day treatment cycles (Cycles 1 to 6) along with an intravenous (IV) infusion of rituximab 375 milligram per square meter (mg/m^2) on Day 1 of Cycle 1 followed by 500 mg/m^2 on Day 1 of each subsequent cycles (Cycles 2 to 6). Cycle duration=28 days. Participants received 6 cycles of chlorambucil plus rituximab or until PD or any other treatment discontinuation criterion was met.
Period: Overall Study
Arm/Group | Acalabrutinib | Chlorambucil Plus Rituximab
Started (Randomized) | 77 | 78
Safety Analysis Set (SAS) (SAS included all participants who received at least 1 dose of study treatment.) | 77 | 73
Completed | 0 | 0
Not Completed | 77 | 78
Not completed — Withdrawal by Subject | 1 | 9
Not completed — Death | 2 | 5
Not completed — Remained on study at time of DCO | 74 | 64

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants.
Groups:
- Acalabrutinib: Participants received acalabrutinib 100 mg orally BID in 28-day cycles until PD or any other treatment discontinuation criterion was met.
- Chlorambucil Plus Rituximab: Participants received chlorambucil 0.5 mg/kg body weight orally on Day 1 and Day 15 of all 28-day treatment cycles (Cycles 1 to 6) along with an IV infusion of rituximab 375 mg/m^2 on Day 1 of Cycle 1 followed by 500 mg/m^2 on Day 1 of each subsequent cycles (Cycles 2 to 6). Cycle duration=28 days. Participants received 6 cycles of chlorambucil plus rituximab or until PD or any other treatment discontinuation criterion was met.
- Total: Total of all reporting groups
Arm/Group | Acalabrutinib | Chlorambucil Plus Rituximab | Total
Number analyzed (Participants) | 77 | 78 | 155
Age, Continuous [Median (Full Range); unit: years] | 64.0 [38 to 86] | 67.0 [21 to 87] | 65.0 [21 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 31 | 65
  Male | 43 | 47 | 90
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 77 | 75 | 152
  White | 0 | 3 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Non-Hispanic or Latino | 77 | 76 | 153

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Assessed by BICR
Description: PFS was defined as the time from randomization to PD (assessed by BICR according to International Workshop on Chronic Lymphocytic Leukaemia [iwCLL] 2018 guideline criteria) or death due to any cause. PD was defined as meeting at least 1 of the below criteria of groups(g) A or B. gA: increase of ≥50% from baseline (BL) or from response in lymph nodes or liver and/or spleen size; any constitutional symptoms; increase of ≥50% over nadir with absolute count ≥ 5×10^9/liter (L) in circulating lymphocyte count (CLC); gB: decrease of ≥50% from BL secondary to CLL in platelet count; decrease of ≥2 gram per deciliter (g/dL) from BL secondary to CLL in hemoglobin (Hb); increase of CLL cells by ≥50% on successive biopsies in bone marrow (BM). Median PFS was calculated using Kaplan-Meier method and its confidence interval (CI) using Brookmeyer-Crowley method.
Time Frame: Response evaluations performed every 12 weeks from Cycle 4 Day 1 to Cycle 25, then every 24 weeks until PD or death, up to DCO date of 03 January 2024 (a maximum of approximately 47.5 months)
Population: FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Acalabrutinib | Chlorambucil Plus Rituximab
Number analyzed (Participants) | 77 | 78
months | NA [NA to NA] — NA indicated that the median, lower and upper limit of 95% CI were not estimable due to insufficient number of participants with events. | 15.54 [11.53 to 17.54]
Statistical Analysis 1: Comparison: Acalabrutinib vs Chlorambucil Plus Rituximab; Test type: Superiority; p < 0.0001, Log Rank; The analysis was performed using the unstratified log-rank test; Hazard Ratio (HR) = 0.08, 95% CI 2-sided [0.03 to 0.18] — HR was calculated using an unstratified Cox model with treatment as the only covariate. The CI for HR was calculated using the profile likelihood method

2. Secondary Outcome: Overall Response Rate (ORR) Assessed by BICR and Investigator
Description: ORR:percentage of participants with complete response(CR),CR with incomplete BM recovery(CRi), partial response(PR)/nodular PR(nPR) assessed by BICR;investigator per IWCLL 2018 criteria at/before initiation of subsequent anti-cancer therapy.CR:No lymph nodes(target lesions)≥1.5 centimeter(cm), spleen<13cm,normal liver;CLC,no constitutional symptoms,platelets≥100,000/microliter(μL),Hb≥11.0 g/dL,BM:normocellular,no CLL cells&B-lymphoid nodules.PR:atleast 2 gA parameters;1 gB parameter need to improve if previously abnormal.If only 1 parameter of both gA,B was abnormal prior to therapy,only 1 needs to improve.gA:Decrease≥50% from BL in lymph nodes,liver & or spleen size,CLC;any constitutional symptoms, gB:platelet≥100,000/μL or increase 50% over BL;Hb≥11g/dL or increase≥50% over BL;BM:presence of CLL cells/B-lymphoid nodules/not done.CRi:all CR criteria+persistent anemia,thrombocytopenia or neutropenia unrelated to CLL,related to drug toxicity.nPR:CR+presence of B-lymphoid nodules in BM.
Time Frame: as for outcome 1
Population: FAS included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Acalabrutinib | Chlorambucil Plus Rituximab
Number analyzed (Participants) | 77 | 78
percentage of participants
  BICR Assessment | 76.6 | 71.8
  Investigator Assessment | 81.8 | 60.3

3. Secondary Outcome: Duration of Response (DOR) Assessed by BICR and Investigator
Description: DOR was defined as the time from response (date of first documented response) to PD or death (absence of PD) as judged by BICR and investigator. PD was defined as meeting at least 1 of the below criteria of group A or group B. Group A: Increase of ≥ 50% from BL or from response in lymph nodes or liver and/or spleen size; any constitutional symptoms; increase of ≥50% over nadir with absolute count ≥ 5×10^9/L in CLC; group B: decrease of ≥50% from BL secondary to CLL in platelet count; decrease of ≥2 g/dL from BL secondary to CLL in hemoglobin; increase of CLL cells by ≥50% on successive biopsies in marrow. Median DOR was calculated using Kaplan-Meier method and its CI using Brookmeyer-Crowley method.
Time Frame: as for outcome 1
Population: FAS included all randomized participants. Only participants with response in each specified category were analyzed in this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Acalabrutinib | Chlorambucil Plus Rituximab
Number analyzed (Participants) | 63 | 56
months
  BICR Assessment: number analyzed (Participants) | 59 | 56
  BICR Assessment | NA [NA to NA] — NA indicated that the median, lower and upper limit of 95% CI were not estimable due to insufficient number of participants with events. | 11.56 [8.28 to 14.26]
  Investigator Assessment: number analyzed (Participants) | 63 | 47
  Investigator Assessment | NA [30.55 to NA] — NA indicated that the median and upper limit of 95% CI were not estimable due to insufficient number of participants with events. | 19.29 [11.47 to NA] — NA indicated that the upper limit of 95% CI was not estimable due to insufficient number of participants with events.

4. Secondary Outcome: Time to Next Treatment (TTNT)
Description: TTNT was defined as the time from the date of randomization to the date of initiation of non-protocol-specified anti-CLL therapy (either medication or radiotherapy for CLL) or death from any cause, whichever occurred first. Median TTNT was calculated using Kaplan-Meier method and its CI was calculated using Brookmeyer-Crowley method.
Time Frame: Response evaluations performed every 12 weeks from Cycle 4 Day 1 to Cycle 25, then every 24 weeks until PD, and survival follow-ups performed every 12 weeks thereafter, up to DCO date of 03 January 2024 (a maximum of approximately 47.5 months)
Population: FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Acalabrutinib | Chlorambucil Plus Rituximab
Number analyzed (Participants) | 77 | 78
months | NA [NA to NA] — NA indicated that the median, lower and upper limit of 95% CI were not estimable due to insufficient number of participants with events. | 26.22 [19.48 to NA] — NA indicated that the upper limit of 95% CI was not estimable due to insufficient number of participants with events.

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization until death due to any cause. The median OS was calculated using Kaplan-Meier method and its CI was calculated using Brookmeyer-Crowley method.
Time Frame: From date of randomization until death due to any cause, up to DCO date of 03 January 2024 (a maximum of approximately 47.5 months)
Population: FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Acalabrutinib | Chlorambucil Plus Rituximab
Number analyzed (Participants) | 77 | 78
months | NA [NA to NA] — NA indicated that the median, lower and upper limit of 95% CI were not estimable due to insufficient number of participants with events. | NA [NA to NA] — NA indicated that the median, lower and upper limit of 95% CI were not estimable due to insufficient number of participants with events.

6. Secondary Outcome: Minimal Residual Disease (MRD) Negativity Rate
Description: The MRD negative rate was defined as the percentage of participants with MRD-negativity (defined as <1 CLL cell per 10,000 leukocytes) measured in the peripheral blood by flow cytometry.
Time Frame: At Cycle 9 (cycle duration: 28 days)
Population: FAS included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Acalabrutinib | Chlorambucil Plus Rituximab
Number analyzed (Participants) | 77 | 78
percentage of participants | 1.3 | 11.5

7. Secondary Outcome: Plasma Concentrations of Acalabrutinib and Its Metabolite ACP-5862
Description: Blood samples were collected to determine the concentration of acalabrutinib and its metabolite ACP-5862 in plasma.
Time Frame: Pre-dose, and at 1, 2, 4 hours post-dose on Day 1 of Cycle 2 (cycle duration: 28 days)
Population: Pharmacokinetic (PK) analysis set included all randomized participants who received at least 1 dose of study drug, for whom there was at least 1 reportable post-dose PK concentration available. Only participants with data collected for each specified timepoints are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Acalabrutinib
Number analyzed (Participants) | 71
nanogram per milliliter
  Acalabrutinib: Pre-dose: number analyzed (Participants) | 62
  Acalabrutinib: Pre-dose | 4.057 (123.8)
  Acalabrutinib: 1 hour post-dose: number analyzed (Participants) | 70
  Acalabrutinib: 1 hour post-dose | 131.941 (424.5)
  Acalabrutinib: 2 hours post-dose | 176.728 (131.9)
  Acalabrutinib: 4 hours post-dose | 56.822 (112.0)
  ACP-5862: Pre-dose: number analyzed (Participants) | 67
  ACP-5862: Pre-dose | 52.314 (60.4)
  ACP-5862: 1 hour post-dose: number analyzed (Participants) | 69
  ACP-5862: 1 hour post-dose | 183.15 (176.1)
  ACP-5862: 2 hours post-dose | 298.758 (102.1)
  ACP-5862: 4 hours post-dose | 222.881 (72.0)

8. Other Pre Specified Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence (other than progression of the malignancy under evaluation) in participant or clinical study participant administered medicinal product and which does not necessarily had a causal relationship with treatment. A serious adverse event (SAE) was an AE occurring during any study phase, that fulfilled 1 or more of following criteria: resulted in death, was life-threatening, required in-participant hospitalization/prolongation of existing hospitalization, resulted in persistent or significant disability or incapacity, was congenital abnormality or birth defect, and was an important medical event that jeopardized participant or required medical treatment to prevent 1 of outcomes listed above. TEAE was any AE that occurred or worsened in severity on or after date of the first dose of study drug up to 30 days after last dose of study drug or prior to initiation of a new anti-CLL therapy, whichever occurred first.
Time Frame: From first dose of study drug (Day 1) up to DCO date of 03 January 2024 (a maximum of approximately 47.5 months)
Population: SAS included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Acalabrutinib | Chlorambucil Plus Rituximab
Number analyzed (Participants) | 77 | 73
Participants
  TEAEs | 74 | 68
  TESAEs | 30 | 17

ADVERSE EVENTS:
Time Frame: From first dose of study drug (Day 1) up to DCO date of 03 January 2024 (a maximum of approximately 47.5 months).
Description: SAS included all participants who received at least 1 dose of study treatment. All-cause mortality was reported in FAS. All participants should receive the same dose within their respective treatment arms.
Groups:
- Chlorambucil Plus Rituximab: Participants received chlorambucil 0.5 mg/kg bodyweight orally on Day 1 and Day 15 of all 28-day treatment cycles (Cycles 1 to 6) along with an IV infusion of rituximab 375 mg/m^2 on Day 1 of Cycle 1 followed by 500 mg/m^2 on Day 1 of each subsequent cycles (Cycles 2 to 6). Cycle duration=28 days. Participants received 6 cycles of chlorambucil plus rituximab or until PD or any other treatment discontinuation criterion was met.
Arm/Group | Acalabrutinib | Chlorambucil Plus Rituximab
All-Cause Mortality (participants affected / at risk) | 2/77 | 5/78
Serious Adverse Events (participants affected / at risk) | 30/77 | 17/73
Other Adverse Events (participants affected / at risk) | 67/77 | 61/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acalabrutinib (N=77) | Chlorambucil Plus Rituximab (N=73)
Pneumonia (Infections and infestations) | 7 (9) | 4 (5)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hepatic enzyme increased (Investigations) | 2 (3) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 1 (1) | 2 (2)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (3)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (2) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 6 (6) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 5 (5) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Central nervous system infection (Infections and infestations) | 1 (1) | 0 (0)
Fournier's gangrene (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acalabrutinib (N=77) | Chlorambucil Plus Rituximab (N=73)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 11 (12)
Upper respiratory tract infection (Infections and infestations) | 9 (13) | 5 (6)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 8 (10)
Alanine aminotransferase increased (Investigations) | 7 (10) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 7 (8) | 2 (3)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 4 (7)
Gamma-glutamyltransferase increased (Investigations) | 5 (6) | 1 (1)
Lymphocyte count increased (Investigations) | 11 (11) | 0 (0)
Neutrophil count decreased (Investigations) | 10 (19) | 18 (32)
Platelet count decreased (Investigations) | 10 (17) | 9 (17)
Weight increased (Investigations) | 10 (10) | 6 (8)
White blood cell count decreased (Investigations) | 0 (0) | 9 (24)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 (5) | 4 (5)
Hyperuricaemia (Metabolism and nutrition disorders) | 9 (13) | 3 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (8) | 5 (6)
Hypophosphataemia (Metabolism and nutrition disorders) | 4 (5) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 9 (13) | 11 (21)
Dizziness (Nervous system disorders) | 9 (13) | 6 (6)
Headache (Nervous system disorders) | 15 (17) | 6 (7)
Petechiae (Skin and subcutaneous tissue disorders) | 4 (6) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 10 (11) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (6) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 12 (14) | 2 (3)
Nausea (Gastrointestinal disorders) | 4 (5) | 3 (3)
Vomiting (Gastrointestinal disorders) | 4 (5) | 3 (4)
Chills (General disorders) | 0 (0) | 7 (9)
Leukocytosis (Blood and lymphatic system disorders) | 11 (12) | 1 (2)
Fatigue (General disorders) | 4 (4) | 3 (3)
Pyrexia (General disorders) | 6 (7) | 6 (6)
COVID-19 (Infections and infestations) | 22 (23) | 10 (10)
Hepatitis B reactivation (Infections and infestations) | 8 (8) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-04-03): https://cdn.clinicaltrials.gov/large-docs/92/NCT04075292/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/92/NCT04075292/SAP_001.pdf